CLINICAL TRIAL: NCT03448432
Title: Prevalence Study of the Etiologies of Pregnancy Anemias
Brief Title: Prevalence Study of the Etiology of Pregnancy Anemia
Acronym: PREGAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PREGAN (29BRC17.0155)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy Anemia
Keywords: Pregnancy Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia during pregnancy occurs in 41% of women. The most common etiology is iron deficiency, but studies to determine prevalence of other causes of anemia in pregnancy are still lacking. However, anemia in pregnancy lead to adverse pregnancy outcomes and increase risk of maternal and fœtal morbidity and mortality. Specific management of anemia is so needed.

ELIGIBILITY:
Inclusion Criteria:

* woman 18-years or older
* woman with a normal pregnancy
* anemia with accidental or symptomatic discovery, whatever the term of pregnancy
* non opposition collected

Exclusion Criteria:

* Refuse to participate
* Stopped pregnancy whatever the term
* Medical abortion of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman with anemia
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-10-27 (Estimated); Study Completion 2019-12-27 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the etiologies of anemias occured during pregnancy | from date of inclusion until 6 weeks after delivery
  Anemia in pregnancy is defined as hemoglobin level (Hb) < 11 g/dL in the first and the third trimesters, and Hb < 10.5 g/dL in the second trimester.

SECONDARY OUTCOMES:
Study of obstetrical complications in women with anemia | from date of inclusion until delivery
  * Measure of the incidence of postpartum haemorrhage, instrumental extractions, caesareans sections, premature delivery, intra-uterine growth restriction or small for gestational age, placenta abruption, preeclampsia and low birth-weight newborn (<3rd and <10th percentile under neonatal morphometry curves)
  * Level of release,
  * 1-, 3- and 5-minutes Apgar score,
  * Arterial ans venous cord potential hydrogen (pH)
Study of the evolution of anemia during pregnancy and postpartum | from date of inclusion until 6 weeks after delivery
  Measure of the Hb level monthly and at 6 weeks after delivery
Describe the etiological and therapeutic management of pregnancy anemias | from date of inclusion until 6 weeks after delivery
  therapeutic management : etiologic treatment (supplemental iron, vitaminic replacement, others) and symptomatic treatment (numbers and rhythm of transfusions)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France